CLINICAL TRIAL: NCT02863237
Title: Predictors of Weaning Outcomes for Brain Injured Patients: a Prospective, Observational Cohort Study
Brief Title: Predictors of Weaning Outcomes for Brain Injured Patients
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: KY2016-018-02
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2018-01

CONDITIONS: Brain Injuries
Keywords: brain injury; mechanical ventilation; weaning
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- weaning failure group: Patients reconnected to the ventilator within 48 hours after SBT will be designated the weaning failure group
- weaning success group: Patients who pass the SBT and breathing without ventilator support within 48 hours are designated the weaning success group

SUMMARY:
Brian injured patients are predisposed to various complications related to mechanical ventilation. Appropriate decision making of the weaning is crucial and validated predictive parameters are desirable. In present study, the investigators aim to a) validate the electrical activity of diaphragm (EAdi) derived parameters, and b) evaluate the traditional predictive parameters in weaning prediction in brain injured patients.

DETAILED DESCRIPTION:
In general intensive care unit (ICU), about 20% patients are ventilated because of neurological illness. This proportion might be much higher in brain injured patients. As with general intensive care patients, brain injured patients are predisposed to a number of complications associated with mechanical ventilation. Both unnecessarily delaying and premature attempts of withdrawal of mechanical ventilation will increase the rate of complications, prolonged mechanical ventilation, the length of stay, motility, and the cost.

Numerous studies had examined factors that predict combined liberation/extubation outcomes, including vital capacity (VC), minute ventilation(VE), and maximum inspiratory pressure (MIP), airway pressure developed 100 ms after the beginning of inspiration against an occluded airway (P0.1), breathing pattern variability (BPV), and the "rapid shallow breathing index" (RSBI, Breathing frequency-tidal volume ratio, f/Vt). The introduction of Neurally Adjusted Ventilatory Assist (NAVA) has made available a standardized and validated method to monitor and measure diaphragm electrical activity (EAdi) both during conventional modes of ventilation and spontaneous breathing trail (SBT). Neuroventilatory efficiency index (NVE, Tidal volume - EAdi ratio, Vt/EAdi) and neuromechanical efficiency index (NME, tidal volume - EAdi ratio, Paw/EAdi) had also been proposed and showed a promising prospect.

However, all those physiological and mechanical parameters are either have limitations on using in brain injured patients, or have not yet been proved to be validity or even had a poor predictive ability. In part this is because respiratory failure of brain injured patient results from two principle etiologic entities: primary pulmonary dysfunction and neurogenic pulmonary dysfunction. The latter brings us quite different characters of brain injury patients, which required specially consideration. Another reason is that, patients with brain injured but no other indication for mechanical ventilation constitute a group in whom the needs for ventilatory support and for an artificial airway might be separate. Previous study that, in neurosurgical patients passed SBT, a median of 2 days elapsed before the attempted extubation, and 45% patients suffered reintubation or tracheostomies. Nonetheless, in most studies, disconnection of ventilatory support and extubation are often lumped together. Although some studies investigated the factors that are predictive of successful extubation, few study considered about the solely liberation of mechanical ventilation.

Therefore, in present study, the investigators separate the liberation of ventilatory support as a standalone part from the traditional weaning/extubation process. Patients are divided into two groups: weaning success and weaning failure, without consideration of the artificial airway status. The primary aims of the study are: a) validate the EAdi derived values, and b) evaluate the traditional predictive parameters in weaning prediction in brain injured patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 80 years
* Mechanical ventilation > 24 hours
* Fulfilling the weaning screen criteria

Exclusion Criteria:

* Moribund or brain dead
* With spinal injury
* Status epilepsy
* Contraindication to EAdi catheter placement
* Severe cardiac disease
* Company with chest or abdominal injury

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brain injured patients receiving mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in Electrical activity of diaphragm measured at the 1, 5, 10, 20, and 30 minutes into the spontaneous breathing trail | 30 minutes
  Measurements are obtained from five consecutive breaths at at the 1, 5, 10, 20, and 30 minutes into the spontaneous breathing trail

SECONDARY OUTCOMES:
Change in Esophageal pressure | 30 minutes
  Measurements are obtained from five consecutive breaths at at the 1, 5, 10, 20, and 30 minutes into the spontaneous breathing trail
Change in Respiratory Rate | 30 minutes
  Measurements are obtained from five consecutive breaths at at the 1, 5, 10, 20, and 30 minutes into the spontaneous breathing trail
Change in Airway pressure | 30 minutes
  Measurements are obtained from five consecutive breaths at at the 1, 5, 10, 20, and 30 minutes into the spontaneous breathing trail
Change in Intrinsic positive end-expiratory pressure | 30 minutes
  Measurements are obtained from five consecutive breaths at at the 1, 5, 10, 20, and 30 minutes into the spontaneous breathing trail
Change in Esophageal pressure time product | 30 minutes
  Measurements are obtained from five consecutive breaths at at the 1, 5, 10, 20, and 30 minutes into the spontaneous breathing trail
Change in Rapid shallow breathing index | 30 minutes
  Measurements are obtained from five consecutive breaths at at the 1, 5, 10, 20, and 30 minutes into the spontaneous breathing trail

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — Beijing Tiantan Hospital
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shi ZH, Jonkman AH, Tuinman PR, Chen GQ, Xu M, Yang YL, Heunks LMA, Zhou JX. Role of a successful spontaneous breathing trial in ventilator liberation in brain-injured patients. Ann Transl Med. 2021 Apr;9(7):548. doi: 10.21037/atm-20-6407. PMID 33987246